CLINICAL TRIAL: NCT00741754
Title: Evaluation of the Unstimulated Whole Saliva Flow During and After Radiotherapy, With the Use of Lauryl-Diethylene-Glycol-Ether Sodium Sulfate Associated With Calcium Hydroxide (hCt20).
Brief Title: Evaluation of the Unstimulated Whole Saliva Flow During and After Radiotherapy, With the Use HcT20
Acronym: EUWSFDAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Éder Ricardo Biasoli, Dental School of University of State of São Paulo - UNESP- Araçatuba
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: upeclin/FOA-Unesp-01; COB-FOA-Unesp-chrishct20
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2009-04-01 (Estimated); Status verified 2008-08

CONDITIONS: Abnormalities, Radiation-Induced
Keywords: salivary flow; oral neoplasm; calcium hydroxide; sodium dodecylsulphate; radiotherapy.
MeSH Terms: conditions — Abnormalities, Radiation-Induced; Mouth Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I, II (Experimental): compare the amount of salivary flow of the same patient at different times.
  Interventions: Other: Mouthrinse with HcT20

INTERVENTIONS:
Other: Mouthrinse with HcT20 — Mouthrinse for 1 minute with 10ml, twice a day. During seven weeks
  Other Names: HcT20

SUMMARY:
The aim of this report was to evaluate the unstimulated whole saliva flow in patients with head and neck cancers during and after the exclusive radiotherapy with an association of lauryl-diethylene-glycol-ether sodium sulfate and calcium hydroxide (Hct20). This study was held at the buccal cancer center of UNESP and involved thirty one patients (n = 31) divided into two groups: Group 1 had seventeen patients (n = 17) submitted to fractioned radiation treatment in the head and neck region at the total dose of 7.000 cGy and had Hct20 during the treatment. Group 2 with fourteen patients (n = 14) started with the use of Hct20 after the end of radiotherapy. A weekly and measured collection of the index of the total non stimulated saliva flow was done on the patients of both groups. The values that were obtained were analyzed statistically through the Bartlett test, the Friedman test and the Wilcox test, to seek an evaluation of effectiveness of the medication on the prevention of the intense drop of the salivary flow during the radiotherapy and do avoid the xerostomia during the post-radiotherapeutic period. The patients from group 1 at the end of the radiotherapy kept the base index of the total non stimulated salivary flow, the ones from group 2 that used the medication association after the radiotherapy had a great improvement of total non stimulated salivary flow and the usage of the Hct20 had a better result on the index of salivary flow during the radiotherapy.

DETAILED DESCRIPTION:
Thirty one patient were observed and treated at Oral Cancer Center - Brazil, between March 1997 and June 2006, distributed into two groups the following way: Group I composed of seventeen patients who utilized Hct20 during the period of the radiotherapy and Group II composed of fourteen patients who utilized the drug association from the radiotherapeutic treatment. The average of the patients in group I was of 58.8 and Group II 64.7 years old. In the distribution, as to sex, group I was composed by fourteen males and three females and in group II 11 male and four female.As to their color, group I presented sixteen white patients and one non-white and group II presented 12 white and two non-white. From the patients in group I, eight referred elitism, six reported social elitism and three denied it; from the patients in group II five referred elitism, two reported social elitism and seven denied it. All the patients, in both groups, presented lesions with primary site in the mouth, oropharynx or larynx with diagnosis of squamous cell carcinoma. The patients included in this research were carriers of oral and oropharynx squamous cell carcinoma guided for exclusive radiotherapeutic treatment.To be accepted in this study, it was established as a requirement that the fields of irradiation included in all occasions the major salivary glands, partially or totally.Patients who used medical drugs wich could interfere in the salivary flow rate, with teeth, mucositis or any other alteration of the oral mucosa after radiotherapy was excluded.Group I was composed of seventeen patients (n=17)that performed eight saliva collection, being one before the treatment (c0) and seven collection (C1to C7) during seven weeks of radiotherapy utilizing Hct20.Group II was composed of fourteen patients (n=14) Who performed nine collections, being one collection (C7) at the end of the treatment without utilizing Hct20, six collections (c8 to C13) utilizing Hct20 the first two months after radiotherapy and two collections (C14 and C15) with three and four months after radiotherapy and after suspending the use of Hct20.The total dose administered to the patients was of 7000 cGy, fractioned in doses of 200 cGy daily, with Five fractions weekly. The composition of Hct20 is 800 ml distilled water, 200 ml of lauryl-diethylene-glycol-ether sodium sulfate (0.125 g/ml) and 2 g of calcium hydroxide.The patients received a vial containing Hct20 and were oriented to perform two oral rinses daily with 10 ml.The collections of unstimulated whole saliva were weekly performed always in the same day of the week, around the same time, before breakfast, without oral hygienization, in the same office with the same illumination and silence and without the presence of companies in the period of the patient in the office.The patients expelled the unstimulated salivary secretion in a test tube calibrated in cubic millimeters with a funnel of eight centimeters of diameter adapted to it.At the end of the collections, wich lasted five minutes, were added three ml of distilled water to each sample, which was stored in a temperature of 6 degree Celsius for 24 hours in order to decrease the bubbles and the foams of the samples. The three ml added to the end of the collection were despised at the moment of the final reading.The values that were obtained were analyzed statistically through the Bartlett test, the Friedman test and the Wilcox test, to seek an evaluation of effectiveness of the medication on the prevention of the intense drop of the salivary flow during the radiotherapy and do avoid the xerostomia during the post-radiotherapeutic period. The patients from group 1 at the end of the radiotherapy kept the base index of the total non stimulated salivary flow, the ones from group 2 that used the medication association after the radiotherapy had a great improvement of total non stimulated salivary flow and the usage of the Hct20 had a better result on the index of salivary flow during the radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* presented lesions with primary site in the mouth, oropharynx or larynx with diagnosis of squamous cell carcinoma.
* the patients were edentulous
* The patients included were guided for exclusive radiotherapeutic treatment.
* To be accepted in this study, it was established as a requirement that the fields of irradiation included in all occasions the major salivary glands, partially or totally.

Exclusion Criteria:

* Patients who used medical drugs wich could interfere in the salivary flow rate, with teeth, mucositis or any other alteration of the oral mucosa after radiotherapy was excluded.

Ages: 40 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-06; Primary Completion 2006-05 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
unstimulated whole saliva flow | ml

CONTACTS AND LOCATIONS:
Overall Officials: Éder Ricardo Biasoli, Principal Investigator — DdS, MsC, PhD. Professor of Oral Diagnosis, School of Dentistry, São Paulo State University - UNESP - Araçatuba - SP - Brazil.
Locations (1):
- Dental School - São Paulo State University, Araçatuba, São Paulo, Brazil

REFERENCES:
- [Result] Larson DL. Long-term effects of radiation therapy in the head and neck. Clin Plast Surg. 1993 Jul;20(3):485-90. PMID 8324987